CLINICAL TRIAL: NCT05538975
Title: Effect of Self-directed and Supervised Pulmonary Rehabilitation Approach on Cough and Sputum Expectoration in Chronic Obstructive Pulmonary Disease
Brief Title: Effect of Self-directed and Supervised Pulmonary Rehabilitation Approach on Cough and Sputum.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afridi Medical Complex (Other)
Responsible Party: Principal Investigator, Usman Farooq, Consultant, Afridi Medical Complex
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0112
Record Dates: First submitted 2022-09-08; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: COPD; Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): home based plan of aerobic exercises, strengthening exercises of upper and lower limbs and huffing and coughing
  Interventions: Other: Physiotherapy Treatment
- Group B (Placebo Comparator): Supervised aerobic exercises, strengthening exercises of upper and lower limbs and huffing and coughing
  Interventions: Other: Physiotherapy Treatment

INTERVENTIONS:
Other: Physiotherapy Treatment — Pulmonary Rehabilitation Techniques

SUMMARY:
Chronic obstructive pulmonary disease (COPD)is a multifactorial, progressive chronic lung disease that causes airflow restriction. Study was conducted To Compare the effects of supervised and self-directed pulmonary rehabilitation on cough and sputum expectoration in patients of chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
To Compare the effects of supervised and self-directed pulmonary rehabilitation on cough and sputum expectoration in patients of chronic obstructive pulmonary disease. It was a randomised control trial and participants were COPD Patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 to 60
* Gender: Both Males & Females.
* Diagnoses with an exacerbation of COPD.
* Informed consent obtained.

Exclusion Criteria:

* Inability to provide informed consent or complete a self-administered questionnaire.
* Patients with trauma.
* Females who were pregnant and breastfeeding.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-08-21 (Actual)

PRIMARY OUTCOMES:
Six minute walk test | 6 months
  to measure distance walked in six minutes
Cough & sputum assessment questionnaire. | 6 months
  recall assesses the frequency and severity of cough and sputum and their impact on everyday life

SECONDARY OUTCOMES:
leicester cough questionnaire | 6 months
  This questionnaire is designed to assess the impact of cough on various aspects of your life.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Alamdar Hussain, Phd, Study Director — Afridi Medical Complex
Locations (1):
- Pulmonary Rehabilitation, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No